CLINICAL TRIAL: NCT06050538
Title: A Prospective Randomized Pilot Study Comparing Transabdominal Properitoneal (TAPP) Versus Totally Extra Peritoneal (TEP) Laparoscopic Inguinal Hernioplasty in Recurrent Inguinal Hernia
Brief Title: Laparscopic Hernioplasty in Recurrent Inguinal Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Islam Hisham, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD.21.03.439
Record Dates: First submitted 2023-08-21; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Recurrent Inguinal Hernia
Keywords: TAPP; TEP; Laparoscopic Inguinal Hernia; Recurrent hernia
MeSH Terms: conditions — Hernia, Inguinal; Hernia | interventions — tetra-4-amidinophenoxypropane; tetraethylpyrazine

STUDY DESIGN:
Intervention Model Description: patients diagnosed with recurrent inguinal hernia. The study population were randomly distributed into 2 groups by computer generating program; group (1) included patients who had Transabdominal preperitoneal (TAPP) approach while group (2) included patients who had Total extraperitoneal (TEP) approach.
Who Masked: Participant, Care Provider
Masking Description: Each patient was randomly allocated to the TAPP group or the TEP group by sequentially numbered, opaque , sealed envelope (SNOSE) technique on the day of surgery. An independent statistician , who was not involved in patient care, generated the randomization sequence via a computer generated random number. The randomization code was contained in opaque sealed envelopes. A junior resident , who opened the envelope , was not actively involved in outcome measurements .Before randomization and during the consent, all patients received an explanation of the objectives of the study, techniques and complications associated with both procedures.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transabdominal preperitoneal (TAPP) (Active Comparator): patients with recurrent inguinal hernia who had Transabdominal preperitoneal (TAPP) approach
  Interventions: Procedure: Transabdominal preperitoneal (TAPP) using polyprolene mesh
- Total extraperitoneal (TEP) approach (Active Comparator): patients with recurrent inguinal hernia who had Total extraperitoneal (TEP) approach
  Interventions: Procedure: Total extraperitoneal (TEP) hernioplasty using polyprolene mesh

INTERVENTIONS:
Procedure: Transabdominal preperitoneal (TAPP) using polyprolene mesh — Transabdominal preperitoneal (TAPP) approach for recurrent inguinal hernia using polyprolene mesh
  Arms: Transabdominal preperitoneal (TAPP)
Procedure: Total extraperitoneal (TEP) hernioplasty using polyprolene mesh — Total extraperitoneal (TEP) approach for recurrent inguinal hernia using polyprolene mesh
  Arms: Total extraperitoneal (TEP) approach

SUMMARY:
The purpose of this study was to compare between laparoscopic transabdominal preperitoneal (TAPP) and totally extraperitoneal (TEP) repair of inguinal hernia in recurrent inguinal hernia.

DETAILED DESCRIPTION:
The primary objective in this study was to compare postoperative pain between the TAPP group and the TEP group. The secondary objective was to compare operative time, intraoperative complications (bleeding, bowel injury, vascular injury), postoperative complications (hematoma, seroma, wound infection), length of hospital stay and recurrence rate with possible risk factors which include gender, age, BMI ,cord lipomas and location of the hernia.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with unilateral or bilateral recurrent inguinal hernias.
* Patients between 18 and 70 years old
* Fit for anesthesia.
* Agree to participate in the study
* Both genders were included.

Exclusion Criteria:

* Unfitness for general anesthesia and operation.
* Age < 18 years or >70 years.
* Complicated hernias (acute irreducible, obstruction or strangulation).
* The presence of mental or psychological disorders.
* Refusal to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 6 months
  by use of visual analog scale (VAS) where (0) refereed to no pain and (10) refereed to the severest pain.

SECONDARY OUTCOMES:
operative time | 6 months
  operative time by minutes was reported to get mean and standard deviation
complications | 6 months
  complications will be described as number and percentages in each group

CONTACTS AND LOCATIONS:
Overall Officials: Islam Hisham, MSc, Principal Investigator — Mansoura University Hospital
Locations (1):
- Mansoura University Hospitl, Al Mansurah, Egypt